CLINICAL TRIAL: NCT04450537
Title: Effects of Anti-JUUL-type Messages on Beliefs, Perceived Harms, and Behavioral Intentions Among Young Adults
Brief Title: PACE Vape Messaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Andrea Villanti, Associate Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00000693; U54DA036114 (NIH)
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Vaping; E-cigarette Use; Electronic Cigarette Use
Keywords: surveys; vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vape Messaging Intervention (Experimental): Participants will be exposed to 10 vape education messages
  Interventions: Behavioral: Vape Messaging Intervention
- Sun Safety Control (No Intervention): Participants will be exposed 10 sun safety messages

INTERVENTIONS:
Behavioral: Vape Messaging Intervention — Participants will be exposed to 10 vape education messages
  Arms: Vape Messaging Intervention

SUMMARY:
The purpose of this study is to examine the effect of exposure to vape education messages on beliefs, perceptions, norms, and behaviors related to electronic vapor product use.

DETAILED DESCRIPTION:
Using content developed from the formative research phase, participants in this randomized controlled trial will either be exposed to ten vape education messages or to ten messages on sun safety, with all messages formatted for social media.

This study will take place over a 1-month period. Individuals who complete the screening survey and are eligible to participate will be invited to complete a 10-15 minute baseline survey at the start of the study. This survey will ask questions about tobacco and electronic vapor product use, and beliefs about and perceptions of vape products. This survey will also ask about exposure to tobacco and e-cigarette marketing, exposure to prevention messaging on vaping and tobacco use, and peer and family influences on tobacco use. During the survey, participants will be presented with and be asked to provide feedback for short health-related messages.

One month after completing this survey, participants will be sent an invitation to the follow-up survey. This survey will again ask about tobacco and electronic vapor product use, and beliefs about and perceptions of vape products.

All study procedures will take place remotely, with surveys conducted online. At the end of the first survey, participants will be eligible to receive a $10 online gift card. Upon completion of the follow-up survey, participants will be eligible to receive a $15 online gift card. In total, participants will be eligible to receive up to $25 for completing both surveys. Those who are ineligible will not be asked to complete the baseline survey and will not be compensated.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-24
* Vermont resident
* Access to a smartphone with internet
* Use of one or more social media site(s) at least weekly

Exclusion Criteria:

* Aged 25 years or older
* Not Vermont resident
* No access to a smartphone with internet
* Use of one or more social media site(s) less than weekly

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 569 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Nicotine/e-cigarette beliefs | Assessed at 1-month follow-up
  True/false/don't know questions about nicotine and electronic vapor/tobacco products
Vape harm perceptions | Assessed at 1-month follow-up
  Harm perception questions about use of electronic vapor/vape products
Vaping-related norms | Assessed at 1-month follow-up
  Questions (5-point Likert scale: 1=Very negative, 5 = Very positive) about others' opinion of using electronic vapor/vape products like JUUL

SECONDARY OUTCOMES:
Behavioral intentions | Assessed at 1-month follow-up
  Questions about intent to use electronic vapor/vape products in the next 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C Villanti, PhD, MPH, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — https://www.pacevt.org